CLINICAL TRIAL: NCT00850018
Title: Neuropsychological Dysfunction and Neuroimaging Abnormalities in Neurologically Intact Adults With Sickle Cell Disease - A Pilot Intervention Study
Brief Title: Examining Cognitive Function and Brain Abnormalities in Adults With Sickle Cell Disease - Pilot Intervention Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Elliott Vichinsky, MD, Children's Hospital of Oakland and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 633; U54HL070587 (NIH); 2U54HL070587 (NIH)
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle Cell Disease; Sickle Cell Anemia; Hemoglobin SS; Hemoglobin SB0
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive monthly blood transfusions.
  Interventions: Procedure: Monthly blood transfusion regimen
- 2 (Active Comparator): Participants will receive usual care.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Procedure: Monthly blood transfusion regimen — Participants will receive blood transfusions at 3- to 4-week intervals for 6 months for the treatment of SCD-related anemia; the total number of transfusions that participants will receive will vary between six and eight.
  Other Names: Chronic transfusion therapy
  Arms: 1
Behavioral: Usual care — Participants will receive usual care for the treatment of SCD.
  Other Names: Standard care alone, guided by disease symptoms.
  Arms: 2

SUMMARY:
Sickle cell disease (SCD), also known as sickle cell anemia, is an inherited blood disease that can cause intense pain episodes and may lead to organ failure. Preliminary studies have shown that adults with SCD may have brain abnormalities that contribute to problems with cognitive functioning, including attention and memory difficulties. This study will use brain magnetic resonance imaging (MRI) and neuropsychological testing to examine the differences in cognitive functioning in adults with SCD who are treated for anemia with monthly blood transfusions for 6 months versus adults with SCD who receive usual care for 6 months.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder. Symptoms include anemia, infections, organ damage, and intense episodes of pain, which are called "sickle cell crises." In the past, SCD was considered a fatal disease, and many people with SCD died at a young age. Due to advances in medical care, people with SCD are now living longer lives; however, they often experience a deterioration in quality of life due to progressive organ failure. Past research has suggested that children with SCD commonly have frontal lobe dysfunction syndrome, which is a brain disorder that can affect cognitive functioning in areas such as attention, concentration, information processing, and decision making. Often times, however, neurocognitive and brain disorders are not diagnosed or treated in people with SCD. In preliminary brain imaging studies, at least half of adult participants with SCD had visible cognitive dysfunction, while participants without SCD rarely had visible changes in the brain. Brain dysfunction may be one of the most important and least-studied problems affecting adults with SCD.

Most people with SCD have anemia, or low levels of red blood cells, which are the cells that carry oxygen to the body's tissues, especially the brain. Research has shown that in people with anemia who do not have SCD, memory and attention problems have decreased after receiving treatment for anemia. The purpose of this study is to determine whether people with SCD who receive monthly blood transfusions to treat their anemia experience greater cognitive functioning than adults with SCD who receive usual care.

The first phase of this study was an observational study that enrolled adults with SCD and a control group of healthy adults who did not have SCD. Study procedures included questionnaires, neuropsychological testing, and MRI testing. At the end of the first phase, participants were asked if they were willing to take part in a second phase of the overall study in the future. Enrollment into the first phase ended in February 2008.

This current pilot study is the second phase of the overall study. In this study, participants will begin by completing questionnaires, a medical history review, a physical exam, a neurological exam, and a blood collection. Women will provide a urine sample for a pregnancy test. An MRI and neuropsychological testing will also occur. Participants will then be randomly assigned to receive either blood transfusions or usual care for 6 months. Participants assigned to blood transfusions will receive the transfusions every 3 to 4 weeks for 6 months. Before each transfusion, participants will undergo blood collection and a review of medical history and medication history. Participants assigned to usual care will receive a telephone call from study researchers at Months 1, 2, 4, and 5, at which time medical and medication history will be reviewed. At study visits at Months 3 and 6, these participants will also undergo a blood collection. At Month 6, all participants will complete health and quality of life questionnaires, neuropsychological testing, and an MRI.

ELIGIBILITY:
Inclusion Criteria:

* Completion of all components of the Phase 1 study (NCT00528801)
* Wechsler Adult Intelligence Scale (WAIS) III-Performance IQ (PIQ) score less than or equal to 90
* Hemoglobin less than or equal to 9.0 g/dL

People who did not complete Phase I of the study are eligible for enrollment in this study if they meet all of the following criteria:

* Capable of giving informed consent for the study
* Willing to undergo transfusion therapy for 6 months
* African descent
* Proficient/fluent in English
* Hemoglobin electrophoresis confirming hemoglobin SS or SB0 (less than or equal to 15%)
* WAIS III-PIQ score less than or equal to 90
* Hemoglobin less than or equal to 9.0 g/dL
* Mini-Mental Status Examination (MMSE) score of greater than or equal to 20
* Profile of Mood States (POMS) score on the Depression-Dejection Subscale less than or equal to 40

Exclusion Criteria:

People who meet any of the following criteria are disqualified from enrollment in this study:

* History of life threatening or serious transfusion complications
* Lack of venous access
* Current enrollment in the Arginine study (NCT00513617)
* Pregnant
* Refusal of transfusion
* History of unexplained severe hemolytic transfusion reaction
* History of serious allergic, pulmonary transfusion reaction requiring hospitalization
* Positive auto-immune hemolytic anemia (direct Coombs test with IgG and complement)
* Multiple (three or more) clinically significant allo-antibodies, due to common antigens (e.g., EC, Kel)
* Uncommon, clinically significant antibody that results in difficulty in finding matched units (e.g., anti-JKB)
* Currently taking Hydroxyurea and not on a stable dose in the 6 months before study entry
* Creatinine level greater than 1.7 mg/dL
* Ferritin level greater than 1,500 ng/mL or quantitative liver iron level greater than 7 mg/g dry weight and not currently on iron chelation therapy. (This is a pilot transfusion in which only 6 months of transfusion will be utilized. The likelihood of iron overload induced toxicity from the transfusions over the 6 months is very small. Furthermore, ferritin is disproportionately elevated in SCD and overestimates the iron burden. Therefore, a quantitative liver iron and/or ferritin level has been included as criteria for exclusion.)
* Major infarct identified on Phase I MRI
* Currently on Procrit or related drug that stimulates red blood cell production

In addition to the exclusion criteria listed above, people who did not complete Phase I (or who completed Phase I more than 1 year prior to enrollment into this study) are disqualified for enrollment in this study if they meet any of the following criteria:

* Overt stroke
* Previous evidence of an abnormal MRI or computed axial tomography (CT) scan other than small periventricular or watershed lesions
* History of head injury that resulted in neurological symptoms or medical visit
* Abnormal neurological exam with focal findings
* Alcohol consumption exceeding 14 drinks/week if female or 21 drinks/week if male
* Drug abuse, as defined as using non-prescribed medication
* History of claustrophobia and/or presence of metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body
* Baseline blood pressure greater than 140/90 mm Hg on two repeated measurements. A second measurement is needed only if the first is greater than 140/90 mm Hg.
* History of uncontrolled hypertension
* Any long-term disorder that may result in neurocognitive or brain dysfunction that is not secondary to SCD, including any of the following:

  * Inflammatory arterial disorders (e.g., lupus, polyarteritis)
  * History of cancer requiring chemotherapy and/or radiation
  * Untreated hyperlipidemia
  * Diabetes
  * Ongoing active infection such as HIV, tuberculosis, or sarcoidosis
  * History of long-term blood transfusion
  * Long-term kidney failure/dialysis
  * Long-term lung disease characterized by a need for oxygen
  * Morbid obesity (i.e., weight greater than 115 kg)
  * Heart disease, including a history of congestive heart failure, history of severe coronary artery disease characterized by angioplasty or surgery, or history of angina
  * Active hepatitis or liver failure
  * Acquired or congenital immune deficiency
  * History of psychoses (e.g., delusions, hallucinations) and/or schizophrenia
  * Neurodegenerative disorder
  * Genetic disorder associated with neurocognitive dysfunction such as Down Syndrome
  * Other long-term illness or disorder other than SCD that will adversely affect the person's performance in the study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2004-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Measured at Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Vichinsky, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (14):
- United States (14):
  - Children's Hospital & Research Center at Oakland, Oakland, California
  - Howard University, Washington D.C., District of Columbia
  - Memorial Cancer Institute, Hollywood, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Johns Hopkins, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute at Wayne State University, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Texas Medical Branch, Galveston, Texas